CLINICAL TRIAL: NCT01931735
Title: Prospective Trial of Arthroscopic Meniscectomy for Degenerative Meniscus Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E0924-R; 1I01RX000924-01A2 (NIH)
Record Dates: First submitted 2013-08-23; First posted 2013-08-29 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Meniscus Tear
Keywords: menisci; tibial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Randomized Meniscectomy (Experimental): This group will have a partial meniscectomy
  Interventions: Procedure: Randomized Meniscectomy
- Randomized Lavage (Active Comparator): This group will have arthroscopy and lavage
  Interventions: Procedure: Randomized Lavage
- Standard of Care Meniscectomy Pre-Amend (Other): Pre-Amendment: surgeons determined standard of care option, meniscectomy, best benefited the patient. Therefore, the patient was not randomized.
  Interventions: Procedure: Standard of Care Meniscectomy Pre-Amend
- Standard of Care Meniscectomy Post-Amend (Other): Post Amendment: patients received a meniscectomy as a standard of care and were observed for 24-months post-operative.
  Interventions: Procedure: Standard of Care Meniscectomy Post-Amend

INTERVENTIONS:
Procedure: Randomized Meniscectomy — Arthroscopic meniscectomy
  Arms: Randomized Meniscectomy
Procedure: Randomized Lavage — Arthroscopic Lavage
  Arms: Randomized Lavage
Procedure: Standard of Care Meniscectomy Pre-Amend — Arthroscopic meniscectomy
  Arms: Standard of Care Meniscectomy Pre-Amend
Procedure: Standard of Care Meniscectomy Post-Amend — Arthroscopic meniscectomy
  Arms: Standard of Care Meniscectomy Post-Amend

SUMMARY:
Arthroscopic meniscectomy is among the most commonly performed orthopedic surgical procedures in the VA system. There remains substantial uncertainty, however, regarding the short term benefits and the long term consequences of arthroscopic meniscectomy in patients with degenerative meniscus tears. Of major concern is the fact that degenerative meniscus tears are associated with osteoarthritis, and it is known that within two years of surgery, arthroscopic debridement for osteoarthritis is no better than placebo in relieving pain and restoring function. Longer term, meniscectomy has been shown to be associated with elevated risk of osteoarthritis development, raising the concern that meniscectomy can actually be harmful. The purpose of this study is to determine whether meniscectomy in the setting of a degenerative meniscus tear is of any clinical value. Determining this would either justify the expenses associated with arthroscopic meniscectomy on a large number of patients, or would identify an area of significant potential cost savings.

DETAILED DESCRIPTION:
The overall goal of this project is to determine whether arthroscopic meniscectomy in degenerative meniscal tears is beneficial from a clinical and scientific viewpoint relative to a non-meniscectomy arthroscopy control. Arthroscopic meniscectomy is among the most commonly performed orthopedic surgical procedures in the VA system and nationally. In the investigators' practice at the VA Palo Alto Healthcare System over the last year, 80% of patients having knee arthroscopy for meniscus tears have been in the 45-70 years age group and 53% of these patients had degenerative meniscal tears without a large unstable flap. these data are comparable to arthroscopic meniscectomy data drawn in other settings. While meniscectomy is a common procedure there remains substantial uncertainty regarding the short term benefits and the long term consequences of arthroscopic meniscectomy in patients with degenerative meniscus tears. Of major concern is the fact that degenerative meniscus tears are associated with osteoarthritis, and it is known that within two years of surgery, arthroscopic debridement for osteoarthritis is no better than placebo in relieving pain and restoring function. Longer term, meniscectomy has been shown to be associated with elevated risk of osteoarthritis development, raising the concern that meniscectomy can actually be harmful. It has also been shown by the group that patients with clinically successful arthroscopic posterior medial meniscectomy have significant change in the rotational motion of the knee during walking. Rotational changes at the knee follow soft tissue damage and have been implicated in the causes for cartilage degeneration.

Thus, there are critical unanswered questions regarding the clinical benefit as well as the scientific basis for arthroscopic meniscectomy for degenerative meniscal tear. To address these questions, this project will conduct a prospective, randomized, blinded, and controlled study of arthroscopic meniscectomy in patients between the ages of 45 and 70 with stable degenerative meniscus tears. In this study, the control group will be a group of patients having arthroscopic lavage of the joint, but no debridement of the stable degenerative meniscus tear. The aims will address clinical (self-reported) and scientific (functional) outcomes of arthroscopic meniscectomy in the time frame lasting up to two years after surgery.

Aim 1: Test the clinical benefit of arthroscopic meniscectomy in the setting of a stable degenerative meniscus tear.

Hypothesis 1a: There will be a significant differences in WOMAC scores between the meniscectomy and the non-meniscectomy/lavage groups at 12 months following surgery.

Hypothesis 1b: The WOMAC scores of the non-meniscectomy/lavage group will not be inferior to the WOMAC scores of the meniscectomy group at 12 months after surgery.

Aim 2: To test the functional effect of arthroscopic meniscectomy in the setting of a degenerative meniscus tear.

Hypothesis 2: Subjects randomized to arthroscopy and meniscectomy will have greater changes in tibio-femoral rotation, knee adduction moment, and knee flexion moment at 12 months following surgery when compared to subjects randomized to arthroscopy and lavage.

In addition to the above principal aims of the study, the investigators will also pursue other exploratory aims:

1. Understand whether arthroscopic meniscectomy for degenerative tear results in accelerated radiographic progression of osteoarthritis (KL score) and regional cartilage thinning (3D MRI thickness maps) relative to a control group.
2. Understand whether tibio-femoral position changes measured in the investigators' gait analysis relate to radiographic progression of osteoarthritis and regional cartilage thinning relative to the control group.
3. Understand whether meniscal tears are associated with activation of the complement system and alteration of gene expression in the synovial lining of the knee, and whether elevated complement activity relates to radiographic OA progression following surgery.
4. Understand whether serum biomarkers are affected in degenerative meniscus tears and whether they will relate to radiographic OA progression or MRI changes following surgery.
5. Investigate whether articular cartilage matrix changes that are measured by advanced MR techniques such as T1rho, sodium, or diffusion MRI can be identified and related to radiographic OA progression or MRI changes following surgery.

This prospective clinical trial with coordinated, multi-disciplinary approach will provide an important clinical and scientific assessment of arthroscopic meniscectomy. It will identify whether surgical treatment is efficacious, an important issue given the costs and risks of surgery. It will also provide new insight into incipient arthritis, yielding information that will impact future patient care.

Update 12/2/2015:

Since the grant was awarded, there has been a growing body of literature published that is directly applicable to the subject of the grant. Specifically, a prospective, randomized study was published in the New England Journal of Medicine in Dec 2013. In that study, the authors did what was proposed in the present study. They found that there was no benefit to meniscectomy in the setting of a degenerative meniscus tear in patients with minimal arthritis of the knee. A very similar study was published a few months before in one of the most important orthopedic journals that focuses on arthroscopy, the American Journal of Sports Medicine. That study was also a prospective randomized study and compared arthroscopic meniscectomy to non-operative treatment for degenerative meniscus tears. The authors of that study also found that arthroscopic meniscectomy for degenerative meniscus tears was of no benefit, this time over non-operative treatment.

When the study was conceived and when the study was funded, there was a genuine uncertainty regarding the appropriate treatment for patients with minimal to no arthritis and a degenerative meniscus tear. With this growing body of literature, however, there is more clarity on this question, and from an ethical standpoint, without genuine equipoise, discussing treatment options and recruiting patients into the study become problematic. The study design was then changed to a prospective observational study of patients with meniscus tears undergoing arthroscopic meniscectomy. The investigators will still be collecting the same data as in the prior randomized trial. The data are patient reported outcome questionnaires, MRI's, and gait analyses at time points from preoperative to two years postoperative. The investigators will also be collecting tissue samples at the time of surgery for the evaluation of inflammatory markers.

Since that time the investigators have reformulated hypotheses. Current aims and hypotheses are:

Aim 1: Determine whether TEAR PATTERN affects PATIENT REPORTED OUTCOMES of arthroscopic meniscectomy Hypothesis 1: There will be greater improvement in patient reported outcomes (WOMET) in patients with displacable meniscus tears than non-displacable meniscus tears.

Aim 2: Determine if STANDARD PREOPERATIVE MR IMAGING can predict PATIENT REPORTED OUTCOME following arthroscopic meniscectomy Hypothesis 2: Patients with MRI evident vertical tears involving 50% of the meniscus or patients with displaced meniscal flaps will have greater improvement in WOMET scores after debridement than those without these MRI findings.

Aim 3: Determine if TEAR PATTERN (and resulting debridement) affects GAIT CHARACTERISTICS at the knee at 12 months post debridement Hypothesis 3: Subjects having debridement of a medial meniscus root tear or a tear that extends through the entire medial meniscus to the periphery will have greater adduction moment and tibial external rotation, and lower flexion angle range of motion than patients who have retention of circumferential fiber continuity or a lateral tear.

Aim 4a: Determine if INFLAMMATORY MARKERS in the synovium at the time of surgery relate to PREOPERATIVE PAIN and PREOPERATIVE MENISCAL TEAR PATTERN.

Hypothesis 4a: Greater inflammation in the synovium will be correlated with greater preoperative pain and with more severe preoperative meniscal damage.

Aim 4b: Determine if INFLAMMATORY MARKERS in the synovium at the time of surgery relate to PATIENT REPORTED OUTCOME following arthroscopic meniscectomy.

Hypothesis 4b: Greater inflammation in the synovium at the time of surgery will be related to greater improvement in pain at three months following surgery.

Aim 5:Determine if PREOPERATIVE GAIT CHARACTERISTICS (knee flexion moment, knee adduction moment, and knee flexion angle) are related to preoperative WOMET scores Hypothesis 5: There will be a negative relationship between WOMET score and knee flexion moment preoperatively.

In addition to the above aims, the investigators will continue to pursue the exploratory aims that were described in the grant application. These are exploratory because they relate to osteoarthritis progression, an outcome that may not be measurable at the one year time frame. The exploratory aims and hypotheses are:

Exploratory Aim 1: Determine if TEAR PATTERN (and subsequent debridement) influences rate of osteoarthritis progression as measured by articular cartilage thinning at 2 years.

Exploratory Hypothesis 1: Tear patterns that involve the meniscal root or complete disruption of the circumferential fibers of the meniscus will exhibit more rapid progression of osteoarthritis than other tear patterns.

Exploratory Aim 2: Determine if GAIT DIFFERENCES (kinematic and kinetics) influence the rate of osteoarthritis progression as measured by articular cartilage thinning at 2 years.

Exploratory Hypothesis 2: Greater adduction moment and external rotation will be related to greater cartilage thinning (2 years - pre operative).

Exploratory Aim 3: Determine if INTRAOPERATIVE SYNOVIAL BIOPSY markers of inflammation are correlated with osteoarthritis progression.

Exploratory Aim 4: Determine if FINDINGS FROM ADVANCED MR IMAGING (T1Rho, Sodium, Diffusion) are correlated with osteoarthritis progression.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age between 45 and 70 years
* Degenerative meniscus tear as seen on standard clinical MRI scan
* Complaint of "mechanical symptoms" which would include popping, catching, or locking of the knee
* Persistent symptoms for a minimum of three months despite conservative management
* Patient is enrolled for arthroscopic meniscectomy
* Subject agrees to the study follow-up schedule and signs informed consent.

Exclusion Criteria:

* Radiographic osteoarthritis of the knee in any compartment greater than KL grade 2
* Prior knee arthroscopy within two years of study enrollment
* Unable to have an MRI scan
* Does not agree to participate

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J. Giori, MD PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edd SN, Giori NJ, Andriacchi TP. The role of inflammation in the initiation of osteoarthritis after meniscal damage. J Biomech. 2015 Jun 1;48(8):1420-6. doi: 10.1016/j.jbiomech.2015.02.035. Epub 2015 Feb 26. PMID 25798759
- [Background] Edd SN, Netravali NA, Favre J, Giori NJ, Andriacchi TP. Alterations in knee kinematics after partial medial meniscectomy are activity dependent. Am J Sports Med. 2015 Jun;43(6):1399-407. doi: 10.1177/0363546515577360. Epub 2015 Mar 31. PMID 25828080

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Meniscectomy: This group will have a partial meniscectomy
  Meniscectomy: Arthroscopic meniscectomy
- Randomized Lavage: This group will have arthroscopy and lavage
  Arthroscopic Lavage: Arthroscopic Lavage
- Standard of Care Meniscectomy Pre-Amendment: Pre-Amendment: surgeons determined standard of care option best benefited the patient.
- Standard of Care Meniscectomy Post Amendment: Post Amendment: patients received a meniscectomy as a standard of care and were observed for 24-months post-operative.
Period: Randomized Phase
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Started | 4 | 3 | 9 | 0
Completed | 2 | 1 | 4 | 0
Not Completed | 2 | 2 | 5 | 0
Not completed — Lost to Follow-up | 2 | 2 | 5 | 0
Period: Observational Non-Randomized Phase
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Started | 2 (Participants continued from the randomized phase) | 1 (Participants continued from the randomized phase) | 0 | 11 (Participants recruited post-amendment)
Completed | 2 | 1 | 0 | 9
Not Completed | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Meniscectomy Pre-Amendment: Pre-Amendment: surgeons determined standard of care option, meniscectomy, best benefited the patient.
- Total: Total of all reporting groups
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment | Total
Number analyzed (Participants) | 4 | 3 | 9 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.5) | 54.3 (3.5) | 55.6 (7.7) | 54.5 (10.8) | 55.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1
  Male | 4 | 2 | 9 | 11 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 2 | 6 | 5 | 14
  Hispanic | 1 | 0 | 1 | 2 | 4
  Unknown | 2 | 0 | 2 | 0 | 4
  African American | 0 | 1 | 0 | 3 | 4
  Other | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 9 | 11 | 27
Total WOMET Score [Mean (Standard Deviation); unit: units on a scale] — Western Ontario Meniscal Evaluation Tool (WOMET) is a standardized and validated survey used to evaluate the pain and function of patients with a degenerative meniscal tear. The survey consists of 16 questions regarding physical symptoms, sports/recreation/work/lifestyle, and emotions. Each question is answered via a visual analog scale (VAS) of 0-100mm for a total score of 1600, where higher numbers are worse. The score is then transformed into a percentage, where 0 is the worst pain and functioning and 100% is no pain and fully functioning.
  units on a scale | 44.8 (31.5) | 45.2 (9.1) | 27.5 (12.2) | 33.1 (22.5) | 34.2 (20.2)
KOOS Pain Score [Mean (Standard Deviation); unit: units on a scale] — Knee injury and Osteoarthritis Outcome Score (KOOS) is a standardized and validated survey used to evaluate the condition of osteoarthritis of the knee. The KOOS Pain scale consists of 9 questions, with each response valued on an ordinal scale of 0-4, and with at total score of 36. Higher numbers indicate more symptoms and physical disabilities. The score is then transformed into a percentage, where 0% is the worst pain and 100% is no pain.
  units on a scale | 29.6 (8.5) | 47.2 (11.78) | 40.1 (12.7) | 42.9 (17.9) | 40.7 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: WOMET Score
Description: Western Ontario Meniscal Evaluation Tool (WOMET) is a standardized and validated survey used to evaluate the pain and function of patients with a degenerative meniscal tear. The survey consists of 16 questions regarding physical symptoms, sports/recreation/work/lifestyle, and emotions. Each question is answered via a visual analog scale (VAS) of 0-100mm for a total score of 1600, where higher numbers are worse. The score is then transformed into a percentage, where 0 is the worst pain and functioning and 100% is no pain and fully functioning.
Time Frame: one year post baseline
Population: Randomize Meniscectomy: 2 lost to follow-up. Randomized Lavage: 2 lost to follow-up. Standard of Care Meniscectomy Pre-Amendment: 5 lost to follow-up. Standard of Care Meniscectomy Post Amendment: 1 withdrew participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Number analyzed (Participants) | 2 | 1 | 4 | 10
units on a scale | 57.5 (42.2) | 99.4 | 37.0 (18.1) | 63.9 (21.9)

2. Primary Outcome: WOMET Score
Description: as for outcome 1
Time Frame: two years post baseline
Population: Randomize meniscectomy: 2 lost to follow-up. Randomized Lavage: 2 lost to follow-up. Standard of care meniscectomy pre-amendment: not in protocol to follow subjects 2 years post baseline. Standard of care meniscectomy post-amendment: 1 withdraw, 1 adverse event.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Number analyzed (Participants) | 2 | 1 | 0 | 9
units on a scale | 49.0 (50.0) | 99.6 |  | 57.4 (27.9)

3. Primary Outcome: Gait Knee Adduction Moment
Description: Knee adduction moment describes the medial/lateral load distribution of the knee measured while walking in a gait laboratory. Before normalization to account for size, the knee adduction moment is expressed in Nm. However, to account for different sized people, the knee adduction moment is transformed and expressed in percentage of body weight times height (%BW*ht). Higher knee adduction moments have been linked to more severe osteoarthritis (OA).
Time Frame: Two year post baseline
Population: Standard of Care Meniscectomy Pre-Amendment group were not assessed for this outcome. Randomized Meniscectomy: 1 was not assessed due to relocation, 2 were lost to follow-up. Randomized lavage: 2 participants were lost to follow-up. Standard of Care Meniscectomy Post Amendment: 1 had an adverse event, 1 participant withdrew from the study.
Measure: Mean (Standard Deviation); unit: percentage of body weight times height
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Number analyzed (Participants) | 1 | 1 | 0 | 9
percentage of body weight times height | -3.32 | -5.40 |  | -2.15 (0.51)

4. Primary Outcome: Average Rotation During Stance
Description: Degree of external tibial rotation averaged over the stance phase of gait.
Time Frame: Two years post baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Number analyzed (Participants) | 1 | 1 | 0 | 8
degrees | 12.5 | 8.2 |  | 8.9 (4.7)

5. Secondary Outcome: KOOS Pain Score
Description: Knee injury and Osteoarthritis Outcome Score (KOOS) is a standardized and validated survey used to evaluate the condition of osteoarthritis of the knee. The KOOS Pain scale consists of 9 questions, with each response valued on an ordinal scale of 0-4, and with at total score of 36. Higher numbers indicate more symptoms and physical disabilities. The score is then transformed into a percentage, where 0% is the worst pain and 100% is no pain.
Time Frame: two years post baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Number analyzed (Participants) | 2 | 1 | 0 | 9
units on a scale | 48.6 (41.2) | 100 |  | 68.5 (26.3)

6. Secondary Outcome: KOOS Pain Score
Description: as for outcome 5
Time Frame: one year post baseline
Population: Randomize meniscectomy: 2 lost to follow-up. Randomized Lavage: 2 lost to follow-up. Standard of care meniscectomy pre-amendment: 5 lost to follow-up. Standard of care meniscectomy post-amendment: 1 withdraw
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Number analyzed (Participants) | 2 | 1 | 4 | 10
units on a scale | 38.9 (39.3) | 100 | 36.8 (15.4) | 66.7 (16.9)

7. Secondary Outcome: TNFa
Description: Tumor necrosis factor-alpha (TNFa) is a pro-inflammatory cytokine that has been linked to the presence of radiographic signs of osteoarthritis (OA), cartilage volume loss over time, increased disease severity, and risk of OA progression. Elevated presence of TNFa can indicate more risk for OA. The unit of measure is pg/mL.
Time Frame: Baseline
Population: No participants were assessed for this measure (data were not collected).
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Randomized Meniscectomy | Randomized Lavage | Standard of Care Meniscectomy Pre-Amendment | Standard of Care Meniscectomy Post Amendment
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/9 | 2/11
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/9 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Meniscectomy (N=4) | Randomized Lavage (N=3) | Standard of Care Meniscectomy Pre-Amendment (N=9) | Standard of Care Meniscectomy Post Amendment (N=11)
Car accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Wrist reconstructed due to a car accident injury. Injury is unrelated to the study.
Diabetic Ulcer (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Diabetic ulcer resulted in toe amputation. This adverse event is unrelated to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Meniscectomy (N=4) | Randomized Lavage (N=3) | Standard of Care Meniscectomy Pre-Amendment (N=9) | Standard of Care Meniscectomy Post Amendment (N=11)
Rheumatoid Arthritis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT01931735/Prot_SAP_001.pdf